CLINICAL TRIAL: NCT04491266
Title: Tolerability and Modulatory Action on Neonatal Gastrointestinal Function and Immunity of the Butyrate Releaser N-(1-carbamoyl-2-phenyl-ethyl) Butyramide as New Component for Infant Formula
Brief Title: Tolerability and Modulatory Action of the Butyrate Releaser N-(1-carbamoyl-2-phenyl-ethyl) Butyramide
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Roberto Berni Canani, Associate Professor, Federico II University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 20-13
Record Dates: First submitted 2020-07-25; First posted 2020-07-29 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Safety Issues

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FBA (Experimental): N-(1-carbamoyl-2-phenyl-ethyl) butyramide (FBA) has been developed.
  Interventions: Dietary Supplement: FBA
- placebo (Placebo Comparator): maltodextrins
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: FBA — N-(1-carbamoyl-2-phenyl-ethyl) butyramide (FBA) has been developed.
  Arms: FBA
Dietary Supplement: placebo — maltodextrins
  Arms: placebo

SUMMARY:
Accumulating evidence is showing that gut microbiota could play a key role in gastrointestinal tract and immune system development and function. Many beneficial effects elicited by gut microbiota are mediated its metabolites. Short chain fatty acids (SCFAs) are major metabolites produced by gut microbiota. Among SCFA, butyrate has emerged as pivotal regulator of many gastrointestinal function and immune system development and function.

Butyrate is produced by intestinal microbial fermentation of resistant starches and dietary fiber. It regulates several beneficial intestinal and extra-intestinal functions, among the first it serves as the primary energy source for the gut epithelium, increases mineral absorption, stimulates proliferation and differentiation of normal colon epithelial cells, improves the gut barrier function by stimulation of the formation of mucin, antimicrobial peptides, and tight-junction proteins, interacts with the immune system and has anti-inflammatory effects.

Butyrate also seems to regulate the expression of antimicrobial peptides in particular upregulating transcription of cathelicidin thanks to his action of histone deacetylase inhibitor and it has been shown to induce human β-defensin 2 (HBD-2) mRNA expression in colonocytes, although there are few publications reporting its regulation of defensins (Berni Canani R et al. W J Gastroenterol. 2011;17(12):1519). Preliminary data showed that breast milk contains butyrate. Butyrate could be an ideal compound for infant formulas for an efficient regulation of a number of protective actions at gastrointestinal tract level and at systemic level.

A new butyrate releaser, useful for all the known applications of butyrate, presenting physiochemical characteristics suitable for easy oral administration (free from unpleasant organoleptic properties of butyrate): N-(1-carbamoyl-2-phenyl-ethyl) butyramide (FBA) has been developed. The molecule is a butyrate amide with the amino acid phenylalanine, solid, odourless, tasteless, stable at gastric pH, and able to release butyrate constantly throughout gastrointestinal tract.

The aim of the study was to evaluate tolerability and safety profile of a nutritional intervention with FBA in formula fed at term neonates. The effects on the expression of innate immunity biomarkers as well as on neonatal gut function were also assessed.

ELIGIBILITY:
Inclusion Criteria:

* otherwise healthy formula fed-neonates
* born at term (>37 gestational age)
* adequate weight for gestational age

Exclusion Criteria:

* twins,
* infants with history of severe asphyxia,
* meconium aspiration syndrome,
* immunodeficiency,
* congenital infections,
* genetic diseases and chromosomal abnormalities,
* malformations,
* insufficient reliability or presence of conditions that made the patient's compliance with the protocol unlikely,
* infants with any other condition which, in the opinion of the Investigator, is likely to interfere with the ability of the infant to ingest food, or the normal growth and development of the infant, or the evaluation of the infant.

In addition, as maternal exclusion factors:

* history of immune diseases,
* tumors,
* infectious or inflammatory diseases that required antibiotic therapy during pregnancy,
* diabetes,
* gestosis,
* dyslipidemia,
* positive vaginal swab for Group B Streptococcus,
* prolonged rupture of membranes.

Max Age: 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2012-01-09 (Actual); Primary Completion 2013-12-31 (Actual); Study Completion 2013-12-31 (Actual)

PRIMARY OUTCOMES:
safety and tolerability: adverse events | up to 28 days
  number and proportion of subjects with adverse events

SECONDARY OUTCOMES:
percentage of subjects with infantile colics | up to 28 days
  rate of subjects with infantile colics
daily number of bowel movements | up to 28 days
  daily number of bowel movements
stool consistency | up to 28 days
  stool consistency
daily number of regurgitation episodes | up to 28 days
  daily number of regurgitation episodes
fecal levels of of β-defensins 2 (HβD-2) | up to 28 days
change of secretory immunoglobulin A (sIgA) | up to 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- University of Naples Federico II, Naples, Italy

IPD SHARING:
Plan to Share IPD: Undecided